CLINICAL TRIAL: NCT03522064
Title: High Dose Testosterone + Carboplatin in Men With Advanced Prostate Cancer
Brief Title: Bipolar Androgen Therapy + Carboplatin in mCRPC
Acronym: HiTeCH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St Vincent's Hospital, Sydney (Other)
Responsible Party: Principal Investigator, Anthony Joshua, FRACP, Principal Investigator, St Vincent's Hospital, Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HiTECH
Record Dates: First submitted 2018-04-17; First posted 2018-05-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Castration-resistant Prostate Cancer; Homologous Recombination Deficiency
Keywords: Castrate-resistant prostate cancer; bipolar androgen therapy; homologous recombination deficiency; BRCA
MeSH Terms: interventions — testosterone enanthate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High dose testosterone + Carbolplatin (Experimental): 500mg IM enanthate every 4 weeks in combination with ongoing LHRH agent (unless post-orchidectomy) plus Carboplatin AUC 5
  Interventions: Drug: Testosterone Enanthate 100 MG/ML Injectable Solution; Drug: Testosterone Enanthate 100 MG/ML Injectable Solution / Carboplatin AUC 5

INTERVENTIONS:
Drug: Testosterone Enanthate 100 MG/ML Injectable Solution — Testosterone Enanthate is the oil-soluble ester of the androgenic hormone testosterone. Testosterone Enanthate is a clear to pale yellow solution for intramuscular injection. Each pre-filled syringe contains 250mg testosterone enanthate/1mL.
  Other Names: Primoteston Depot
Drug: Testosterone Enanthate 100 MG/ML Injectable Solution / Carboplatin AUC 5 — Testosterone Enanthate is the oil-soluble ester of the androgenic hormone testosterone. Testosterone Enanthate is a clear to pale yellow solution for intramuscular injection. Each pre-filled syringe contains 250mg testosterone enanthate/1mL. Carboplatin as per standard procedures

SUMMARY:
The purpose of this study is to determine the efficacy of BAT and carboplatin in men with metastatic castrate-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
Androgen deprivation therapy (ADT) remains the mainstay of prostate cancer treatment. Though an effective therapy initially, the side effects of ADT are numerous and treatment resistance is inevitable. Castrate-refractory prostate cancer (CRPC) progresses via adaptive mechanisms that allow ongoing androgen receptor (AR) signalling despite castrate levels of androgens.

The concept of cycling between supra- and sub physiological levels of testosterone has been tested recently in studies of "bipolar androgen therapy" (BAT) in which patients are given high dose testosterone in combination with androgen deprivation therapy (ADT) via an LHRH agonist/antagonist. Studies of BAT using IM testosterone have been promising both in terms of PSA responses and quality of life improvements. Additionally, these early phase studies suggest the potential for re-sensitisation to novel anti-androgen therapies.

Though responses have been positive in these early studies a proportion of men fail to respond and data to guide patient selection is lacking. There are data to suggest that patients with DNA repair deficits may be particularly responsive to BAT. Whether these changes serve as predictors of response is unknown as the effect of BAT on the tumour, its microenvironment and peripheral circulating tumour DNA has not been studied in detail. Information on treatment effects may be key to appropriate patient selection for this treatment.

The aim of this study is to assess based on the pre-clinical studies, the combination with carboplatin

ELIGIBILITY:
Inclusion Criteria:

1. Males with histologically confirmed adenocarcinoma of the prostate
2. Confirmed HRD (Homologous recombination defect) in germline and/or somatic DNA analysis (tumour or blood), by a validated assay (see Appendix 1). Mutations in HR genes not listed in appendix 1 will be considered in literature suggests pathogenicity. A maximum of 10 uncharacterised or heterozygous mutations will be included.
3. Age ≥ 18 years
4. ECOG performance status ≤ 1
5. Rising PSA confirmed on two sequential tests ≥1 week apart and a minimum value of 2 ug/L despite castrate levels of testosterone
6. Serum testosterone < 1.7 nmol/L and on an LHRH agent or post orchidectomy ≥ 1 year.
7. Washout of ≥ 4 weeks from prior line of treatment, radiotherapy or surgery (aside from LHRH agent)
8. Adequate bone marrow function (platelets > 100 x 109/L, ANC > 1.5 x 109/L, Hb >100)
9. Adequate liver function (ALT/AST < 1.5 x ULN, bilirubin < 2 x ULN)
10. Adequate renal function (creatinine clearance > 50 ml/min)
11. Adequate cardiac function and reserve after cardiology assessment
12. Archived tissue sample available or willingness to undergo fresh biopsy
13. Willing and able to comply with all study requirements, including treatment, timing and/or nature of required assessments
14. Signed, written informed consent

Exclusion Criteria:

1. Contraindications to investigational product
2. Pain due to metastatic prostate cancer requiring opioid analgesics
3. Evidence of disease progression in sites or extent that, in the opinion of the investigator, would put the patient at risk from testosterone therapy and its potential for initial tumour flare (eg: femoral metastasis at risk of fracture, ureteric obstruction due to nodal disease or cord compression due to spinal metastases).
4. Previous treatment with platinum chemotherapy and/or a PARP inhibitor. However up to 8 men with prior treatment to these agents will be included as an exploratory cohort.
5. Life expectancy of less than 3 months.
6. Brain metastases or leptomeningeal disease
7. History of thromboembolic event and not currently on anticoagulation
8. Prior myocardial infarction or unstable angina within 2 years of study entry
9. Haematocrit ≥ 50%, untreated severe obstructive sleep apnoea or poorly controlled heart failure (NYHA >1)
10. History of another malignancy within 5 years prior to registration. Patients with a past history of adequately treated carcinoma-in-situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or superficial transitional cell carcinoma of the bladder are eligible. Patients with a history of other malignancies are eligible if they have been continuously disease free for at least 5 years after definitive primary treatment.
11. Concurrent illness, including severe infection that may jeopardize the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety.
12. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
PSA Response Rate | 1 year
  >/= 50% fall from baseline PSA

SECONDARY OUTCOMES:
Time to PSA progression | 1 year
  Time to increase in PSA >/=25% from baseline or nadir confirmed on subsequent test >1 week later
Radiological Response Rate | 1 year
  RECIST or PCWG3 Criteria
Safety and Tolerability (Frequency of adverse events as assessed by NCI CTCAE v4.0) | 1 year
  Frequency of adverse events as assessed by NCI CTCAE v4.0

OTHER OUTCOMES:
Changes in ctDNA expression from baseline | 1 year
  Exploratory
Change in serum testosterone and oestradiol levels | 1 year
  Change in serum levels from baseline to Days 14 and 28 of cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Anthony M Joshua, MBBS, PhD, FRACP, Principal Investigator — St Vincent's Hospital
Locations (1):
- Kinghorn Cancer Centre, St. Vincent's Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teply BA, Wang H, Luber B, Sullivan R, Rifkind I, Bruns A, Spitz A, DeCarli M, Sinibaldi V, Pratz CF, Lu C, Silberstein JL, Luo J, Schweizer MT, Drake CG, Carducci MA, Paller CJ, Antonarakis ES, Eisenberger MA, Denmeade SR. Bipolar androgen therapy in men with metastatic castration-resistant prostate cancer after progression on enzalutamide: an open-label, phase 2, multicohort study. Lancet Oncol. 2018 Jan;19(1):76-86. doi: 10.1016/S1470-2045(17)30906-3. Epub 2017 Dec 14. PMID 29248236
- [Background] Schweizer MT, Wang H, Luber B, Nadal R, Spitz A, Rosen DM, Cao H, Antonarakis ES, Eisenberger MA, Carducci MA, Paller C, Denmeade SR. Bipolar Androgen Therapy for Men With Androgen Ablation Naive Prostate Cancer: Results From the Phase II BATMAN Study. Prostate. 2016 Sep;76(13):1218-26. doi: 10.1002/pros.23209. Epub 2016 Jun 24. PMID 27338150
- [Derived] Maia MC, Salgia M, Pal SK. Harnessing cell-free DNA: plasma circulating tumour DNA for liquid biopsy in genitourinary cancers. Nat Rev Urol. 2020 May;17(5):271-291. doi: 10.1038/s41585-020-0297-9. Epub 2020 Mar 17. PMID 32203306